CLINICAL TRIAL: NCT03450655
Title: Cardio Training of Older Adults With Central Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Anna Nordström, Adjunct Professor, Region Västerbotten
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCC-LIFE-4
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Visceral Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Data Analyst will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Weeks 1-10: exercise program in group. Weeks 11-20: no intervention. Weeks 21-31: no intervention.
  Interventions: Other: 10-week aerobic exercise program
- Control group (Experimental): Weeks 1-10: no intervention. Weeks 11-20: no intervention. Weeks 21-31: exercise program at home.
  Interventions: Other: 10-week aerobic exercise program

INTERVENTIONS:
Other: 10-week aerobic exercise program — An aerobic exercise program consisting of 45-60 minute sessions 3 times a week for 10 weeks.

SUMMARY:
Given the increasing prevalence of obesity, there is an urgent need to find better strategies to promote physical activity in the community. The present study will invite 70-year-olds with central (abdominal) obesity to participate in a 10-week aerobic exercise program. Participants will be randomly assigned to one of two equally large groups. The first group will complete the exercise program in instructor-led groups. The second group will complete the program at home with the help of an on-line video.

DETAILED DESCRIPTION:
Central obesity means having a lot visceral fat, that is, fat located in the abdominal cavity. Visceral fat is a well-established risk factor for cardiovascular disease and all-cause mortality.

Participants will be recruited from the Healthy Ageing Initiative (HAI), an ongoing population-based study that invites all 70-year-olds in Umeå, Sweden, to a health examination. The exercise program will focus is on station-based aerobic exercises and resistance exercises, predominantly with participants' own body weight as resistance. The program is progressive, starting at a moderate pace so that participants learn to perform the exercises properly. The intensity will be aimed at 60-80% of maximal exhaustion, and each exercise bout will last 60 seconds with 20 seconds of rest between bouts. The program was developed by seniors in the bachelor's program in exercise physiology at Umeå University, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Healthy Ageing Initiative (a population-based intervention study in Umeå, Sweden)
* Visceral adipose tissue mass >1 kg (women) or >2 kg (men)

Exclusion Criteria:

* Physical disability that affects ability to perform the exercises
* Heart failure or severe degenerative condition (e.g. malignant cancer or multiple sclerosis)
* Myocardial infarction or stroke in the past year
* Heart condition that can worsen with aerobic exercise (e.g. angina)

Ages: 70 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-09-28 (Estimated); Study Completion 2018-09-28 (Estimated)

PRIMARY OUTCOMES:
Change in visceral adipose tissue mass | 0, 10, 20, and 31 weeks
  Mass (g) measured using Lunar iDXA with CoreScan application (GE Healthcare, Wauwatosa, WI, USA).

SECONDARY OUTCOMES:
Change in body composition | 0, 10, 20, and 31 weeks
  Mass (g) measured using Lunar iDXA with CoreScan application (GE Healthcare, Wauwatosa, WI, USA)
Change in Body Mass Index (kg/m^2) | 0, 10, 20, and 31 weeks
Change in blood pressure (mmHg) | 0, 10, 20, and 31 weeks
  Taken after 15 min of rest
Change in blood-lipid profile | 0, 10, 20, and 31 weeks
Change in fasting blood glucose | 0, 10, 20, and 31 weeks
  Veinous blood samples taken after > 4 h of fasting
Change in isometric muscle strength | 0, 10, 20, and 31 weeks
  Measured in non-dominant hand with dynamometer (Jamar, Lafayette Instrument, USA). The better of two successive trials will be recorded.
Change in physical capacity | 0, 10, 20, and 31 weeks
  Measured using Åstrands Submaximal Test, performed on an electrically braked ergometer bicycle
Change in resting metabolic rate | 0, 10, 20, and 31 weeks
  As measured by indirect calorimetry
Change in health-related quality of life | 0, 10, 20, and 31 weeks
  As measured by RAND-36
Change in self-reported physical activity | 0, 10, 20, and 31 weeks
  Assessed using IPAQ-SF
Change in Microbiota composition | 0, 10, 20, and 31 weeks
  Fecal samples are taken and bacterial DNA is sequenced to determine bacterial composition
Change in dietary habits | 0, 10, 20, and 31 weeks
  85 item food frequency questionnaire
Change in concentration of inflammatory markers | 0, 10, 20, and 31 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nordström, PhD, Principal Investigator — Umeå University
Locations (1):
- Livsmedicin (LIFE), Umeå, Västerbotten County, Sweden

REFERENCES:
- [Derived] Ballin M, Hult A, Bjork S, Lundberg E, Nordstrom P, Nordstrom A. Web-based exercise versus supervised exercise for decreasing visceral adipose tissue in older adults with central obesity: a randomized controlled trial. BMC Geriatr. 2020 May 12;20(1):173. doi: 10.1186/s12877-020-01577-w. PMID 32398024
- [Derived] Ballin M, Lundberg E, Sorlen N, Nordstrom P, Hult A, Nordstrom A. Effects of interval training on quality of life and cardiometabolic risk markers in older adults: a randomized controlled trial. Clin Interv Aging. 2019 Sep 4;14:1589-1599. doi: 10.2147/CIA.S213133. eCollection 2019. PMID 31564841
- [Derived] Ballin M, Lundberg E, Sorlen N, Nordstrom P, Hult A, Nordstrom A. Effects of Interval Training on Visceral Adipose Tissue in Centrally Obese 70-Year-Old Individuals: A Randomized Controlled Trial. J Am Geriatr Soc. 2019 Aug;67(8):1625-1631. doi: 10.1111/jgs.15919. Epub 2019 Apr 23. PMID 31012497

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT03450655/Prot_SAP_000.pdf